CLINICAL TRIAL: NCT03414736
Title: A Randomized, Comparative, Open Label Study to Assess the Safety and Tolerability of 3-arm, Parallel, Repeated Subcutaneous Dose Regimens of SAR425899 in Overweight to Obese Subjects and T2DM Patients Not Requiring Anti-diabetic Pharmacotherapy, With an Optional 6-month Safety Extension Period
Brief Title: A Study on Safety and Tolerability of SAR425899 in Overweight to Obese Subjects and Type 2 Diabetes Mellitus Patients Not Requiring Anti-Diabetic Pharmacotherapy With an Optional 6-month Safety Extension Period
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TDR15516; U1111-1205-1368 (Other: UTN)
Record Dates: First submitted 2018-01-17; First posted 2018-01-30 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — SAR425899

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Daily dose escalation (click-by-click): Starting at dose 1 in the morning with daily increments to dose 2. During the escalation phase, the dose will only be increased if the patient is feeling fine.
  Interventions: Drug: SAR425899
- Cohort 2 (Experimental): Weekly dose escalation in 6 escalation steps (7 dose levels): Starting at dose 1 injected in the morning with weekly increments to dose 2. In case a dose level is not well tolerated by a patient, the treatment should continue at the same dose level for another 7 days before the next dose escalation.
  Interventions: Drug: SAR425899
- Cohort 3 (Experimental): Weekly dose escalation in 4 escalation steps (5 dose levels): Starting at dose 3 with weekly increments to dose 2. In case a dose level is not well tolerated by a patient, the treatment should continue at the same dose level for another 7 days before the next dose escalation.
  Interventions: Drug: SAR425899

INTERVENTIONS:
Drug: SAR425899 — Pharmaceutical form: Solution
  Route of administration: Subcutaneous

SUMMARY:
Primary Objectives:

* Main study: To assess in overweight to obese subjects and type 2 diabetes mellitus (T2DM) patients not requiring anti-diabetic pharmacotherapy the safety and tolerability of 3 different dose escalation regimens of SAR425899 in terms of the relative and absolute frequency and severity of gastrointestinal (GI) adverse events (AEs).
* Six-month safety extension period: To assess the safety and tolerability of SAR425899 after 6 months treatment at the maximum dose that was individually well tolerated during the main part of the study in terms of the relative and absolute frequency and severity of GI AEs.

Secondary Objectives:

Main study and 6-month study extension period:

To assess in overweight to obese subjects and T2DM patients not requiring anti-diabetic pharmacotherapy:

* The effect of once-daily dosing of SAR425899 on body weight (BW), fasting plasma glucose (FPG), and hemoglobin A1c (HbA1c).
* Safety and tolerability.

DETAILED DESCRIPTION:
Main study: The maximum study duration is approximately 12 weeks per patient (up-to 3-week screening period, 8-week treatment period, 3-day post treatment follow-up period).

Six-month study extension period: The maximum study duration is approximately 9 months (up-to 3-week screening period, 8-month treatment period, 3-day post treatment follow-up period).

ELIGIBILITY:
Inclusion criteria:

* Male or female overweight to obese subjects and type 2 diabetes mellitus (T2DM) patients not requiring anti-diabetic pharmacotherapy.
* Patients who are motivated to lose weight.

Exclusion criteria:

* Type 1 diabetes mellitus.
* Body mass index <27 kg/m2.
* Screening hemoglobin A1c (HbA1c; glycosylated hemoglobin) >7.0%.
* Previous treatment with glucose-lowering agent(s) (eg, insulin, thiazolidinediones, metformin, DPP-IV inhibitors (dipeptidylpeptidase 4), SGLT-2 (sodium dependent glucose transporter-2) inhibitors, etc) within the last 6 months.
* Previous treatment with glucagon-like peptide 1 (GLP-1) receptor agonists within the last 6 months.
* Uncontrolled hypertension.
* Laboratory findings at the time of screening: amylase and/or lipase >2 times the upper limit of the normal laboratory range (ULN), alanine aminotransferase >1.5 ULN, total bilirubin >1.5 ULN, serum creatinine levels ≥1.5 mg/dL [males]. ≥1.4 mg/dL [females], screening calcitonin ≥20 pmol/m, fasting serum triglycerides >400 mg/dL.
* Personal or immediate family history of medullary thyroid cancer (MTC) or genetic conditions that predispose to MTC.
* History of weight loss surgery.
* History of pancreatitis or pancreatectomy.
* Pregnant or lactating women.
* Women of childbearing potential (WOCBP) not protected by highly-effective method(s) of birth control and/or who are unwilling or unable to be tested for pregnancy.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2018-10-05 (Actual)

PRIMARY OUTCOMES:
Frequency of gastrointestinal (GI) adverse events (AEs) | Main study: Up to week 8; Six-month study extension period: Up to month 8
  Relative frequency of GI AEs
Frequency of GI AEs | Main study: Up to week 8; Six-month study extension period: Up to month 8
  Absolute frequency of GI AEs
Frequency of GI AEs | Main study: Up to week 8; Six-month study extension period: Up to month 8
  Severity of GI AEs

SECONDARY OUTCOMES:
Change in body weight | Main study: Baseline (D1) to week 8; Six-month study extension period: Baseline (D1) up to month 8
  Change in body weight from baseline to week 8 for the main study and from baseline to month 8 for the study extension period.
Change in fasting plasma glucose (FPG) | Main study: Baseline (D1) to week 8; Six-month study extension period: Baseline (D1) up to month 8
  Change in FPG from baseline to week 8 for the main study and from baseline to month 8 for the study extension period.
Change in hemoglobin A1c (HbA1c) | Main study: Baseline (D1) to week 8; Six-month study extension period: Baseline (D1) up to month 8
  Change in HbA1c from baseline to week 8 for the main study and from baseline to month 8 for the study extension period.
Adverse events (AEs) | Main study: up to week 8; Six-month extension period: up to month 8
  Number of AEs

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (3):
- United States (3):
  - Investigational Site Number 8400002, Saint Paul, Minnesota
  - Investigational Site Number 8400003, Knoxville, Tennessee
  - Investigational Site Number 8400001, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org